CLINICAL TRIAL: NCT00618475
Title: Cognitive Behavioral Treatment of Depression in ESRD Patients on Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: K23DK076980 (NIH); K23DK076980 (NIH)
Record Dates: First submitted 2008-02-15; First posted 2008-02-20 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: End Stage Renal Disease; Depression
Keywords: Depression; End Stage Renal Disease; Kidney Disease; Mental Health
MeSH Terms: conditions — Kidney Failure, Chronic; Depression; Kidney Diseases; Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Individual cognitive behavioral therapy (CBT)
  Interventions: Behavioral: Cognitive behavioral therapy
- Wait-list control (Other): Individual cognitive behavioral therapy (CBT) after 3 month wait-list period
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — 10 sessions
  1 hour per week

SUMMARY:
Depression is second in frequency only to hypertension as a comorbid condition for End Stage Renal Disease (ESRD) patients. The presence of depression has been linked to lower quality of life, more medical comorbidities and shorter lifespan. This project represents the first known attempt at a standardized intervention for depression in ethnically diverse ESRD patients. The study will be conducted at the Parkside Center for Dialysis. Patients will be randomly selected for screening until 80 subjects meet entry criteria and agree to be randomized. Once subjects are screened and enrolled in the study they are randomly assigned to either a treatment or wait-list control condition. After 3 months, the intervention will be completed and both groups will be reassessed. After an additional 3 months, both groups will have received the intervention and pre and post measures for both groups will be available as well as 3 month follow-up for the 1st intervention group.

The following measures will be collected: to obtain a full DSM-IV diagnosis the SCID I and SCID II will be utilized. The BDI will provide a self-report measure of depression. The Hospital Anxiety and Depression Scale (HADS), a measure designed specifically for medically ill patients, will also be administered. Additionally, the Young Schema Questionnaire, a measure which seeks to identify maladaptive (both depressive and anxious) cognitive styles, will be administered. A quality of life measure designed specifically for dialysis patients (KDQOL-SF) will also be given as a means of measuring patient's overall coping and functioning. To better understand the patient's perceptions of their health and illness the Illness Effects Questionnaire will be administered. A demographic information sheet will be completed by the subject in which personal, ethnic, and illness information is collected. Detailed information about the subject's mental health history and treatment as well as current medications will be gathered. Data from routine dialysis laboratories (hemoglobin, creatinine, albumin, Kt/V) will be extracted from the chart.

The intervention will take place in individual format while the subjects are being dialyzed. The intervention will be 10 sixty minute -long weekly sessions spread over not more than 3 months. It will include both cognitive and behavioral skills focused on alleviating depressive affect and identifying maladaptive patterns of thought and behavior. This study would lay the groundwork for future clinical research by helping to develop a culturally competent clinical intervention and demonstrate the feasibility and effectiveness of adapting psychosocial intervention for a medically complex culturally diverse population.

ELIGIBILITY:
Inclusion Criteria:

- hemodialysis patient Depression diagnosis

Exclusion Criteria:

(1) presence of current organic mental disorder (2) schizophrenia (3) bipolar disorder (4) depression with psychotic features (5) current substance abuse or dependence (6) active suicidal intent or plan (7) active homicidal ideation, intent, or plan -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | baseline, completion, 3 month follow-up

SECONDARY OUTCOMES:
Quality of Life | baseline, completion, 3 month follow-up
Clinical biomarkers | baseline, completion, 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cukor, PhD., Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- Parkside Hemodialysis, Brooklyn, New York, United States

REFERENCES:
- [Result] Cukor D, Ver Halen N, Asher DR, Coplan JD, Weedon J, Wyka KE, Saggi SJ, Kimmel PL. Psychosocial intervention improves depression, quality of life, and fluid adherence in hemodialysis. J Am Soc Nephrol. 2014 Jan;25(1):196-206. doi: 10.1681/ASN.2012111134. Epub 2013 Oct 10. PMID 24115478